CLINICAL TRIAL: NCT01947660
Title: Continuous Regional Anesthesia for Septic Limb Orthopedic Surgery
Acronym: ACOSM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5492
Record Dates: First submitted 2013-09-17; First posted 2013-09-20 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2013-09

CONDITIONS: Osteo Arthritis; Cellulitis
MeSH Terms: conditions — Cellulitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous regional anesthesia (Experimental)
  Interventions: Drug: Systemic analgesia + Continuous regional anesthesia
- Systemic analgesia (Active Comparator)
  Interventions: Drug: Systemic analgesia

INTERVENTIONS:
Drug: Systemic analgesia + Continuous regional anesthesia — Systemic analgesia + Continuous regional anesthesia, peri neural for the 2 to 4 first days post-operative
  Arms: Continuous regional anesthesia
Drug: Systemic analgesia — Systemic analgesia as usual
  Arms: Systemic analgesia

SUMMARY:
This study aims to assess the safety of using continuous regional anesthesia for post-operative analgesia during septic limb orthopedic surgery.

The study hypothesis is that continuous regional anesthesia would not induce septic complication in the operated limb and could improve post-operative recovery.

ELIGIBILITY:
Inclusion Criteria:

* Osteo arthritis or cellulitis requiring surgical intervention
* anatomical possibility of regional anesthesia
* age >18 ans
* written informed consent

Exclusion Criteria:

* loco-regional anesthesia impossibility (puncture zone infection, local anesthesics allergie, amiodarone or mexilétine treatment, neurologic deficit for exemple)
* patient under tutelle or curatelle
* pregnant or beast feeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Septic complication in the operated limb | 28 days
  Septic complication in the operated limb Pain score Nausea and vomiting

CONTACTS AND LOCATIONS:
Locations (1):
- CCOM, Illkirch-Graffenstaden, Alsace, France